CLINICAL TRIAL: NCT02707055
Title: A Novel Compound for Alcoholism Treatment: A Translational Strategy - Part II
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination of the study due to the COVID-19 pandemic
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Rhode Island (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 160080; 16-DA-0080
Record Dates: First submitted 2016-03-11; First posted 2016-03-14 (Estimated); Results first posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-10

CONDITIONS: Alcoholism
Keywords: Alcohol Consumption; Alcohol Treatment; Alcoholism; Ghrelin; Ghrelin Antagonism
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — PF-5190457

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-05190457, then placebo (Experimental): Participants with alcohol use disorder received PF-05190457 100 mg twice a day for a maximum of 14 days followed by a minimum of 2-day washout period, then placebo twice a day for a maximum of 14 days.
  Interventions: Drug: PF-05190457; Other: Placebo
- Placebo, then PF-05190457 (Placebo Comparator): Participants with alcohol use disorder received placebo twice a day for a maximum of 14 days followed by a minimum of 2-day washout period then PF-05190457 100 mg twice a day for a maximum of 14 days.
  Interventions: Drug: PF-05190457; Other: Placebo

INTERVENTIONS:
Drug: PF-05190457 — Ghrelin Receptor Inverse Agonist
Other: Placebo — Placebo

SUMMARY:
Background:

Hormones are naturally occurring chemicals in the body. Ghrelin is a hormone that stimulates appetite. It may also stimulate alcohol cravings and use. Researchers want to learn more about alcohol cravings and test if a drug that blocks ghrelin lowers alcohol cravings.

Objective:

To test if the drug PF-05190457 decreases alcohol craving.

Eligibility:

People ages 18-70 who have:

Alcohol use disorder

No other serious medical problems

Woman must be postmenopausal or have had surgery to prevent pregnancy.

Design:

Participants will stay on the inpatient unit here at the Clinical Center for two 2-week stages, which will be separated by at least 2 days. The inpatient phase include:

Taking the study drug or placebo by mouth twice daily

Blood tests

Tasting several sweet solutions

Physical exams

Exposure to alcohol, water, and food cues in a bar-like room. Participants answer questions on a computer.

Blood pressure and heart rate are monitored through an arm cuff and sensors on the chest.

MRIs: Participants lie on a table that slides in and out of the cylinder, and a coil is placed over the head.

They complete tasks on a computer screen while in the cylinder. This lasts up to 2 hours.

Wearing a virtual reality headset, walking around a virtual room, and selecting virtual food and drink.

Physical exams

DETAILED DESCRIPTION:
Objective:

Ghrelin is a 28-amino acid peptide that stimulates appetite and food intake. It is an endogenous ligand for the growth hormone secretagogue receptor (GHSR1a). Preclinical studies suggest that ghrelin modulates alcohol reward processing. Previous work from our research team, indicated that intravenous (IV) ghrelin administration, compared to placebo, results in an acute increase in alcohol craving during a cue-reactivity experiment in alcoholic individuals. Therefore, an oral bioavailable, ghrelin receptor antagonist that is able to pass through the blood brain barrier holds particular promise as a treatment for alcohol use disorder (AUD). This protocol is part of a grant project funded by National Center for Advancing Translational Sciences (NCATS) aimed to generate preliminary evidence in AUD on the safety and efficacy of a ghrelin receptor (GHSR1a) antagonist, PF-05190457, an existing molecule available under the NIH-Industry Pilot Program at NCATS. Completed preclinical and clinical (Protocol #14-AA-0042) work has demonstrated the safety of PF-05190457/alcohol interaction. The goal of this protocol is to conduct a proof-of-concept human laboratory study to assess an early-signal of efficacy of PF-05190457 in AUD.

Study population:

The study population will be AUD individuals (n = 55).

Study Design:

A within-subject, counterbalanced, double-blind, placebo-controlled study.

Outcome measures:

The primary aim will be to determine whether PF-05190457, compared to placebo, reduces alcohol cue-elicited craving. As another outcome will be to determine whether PF-05190457, compared to placebo, reduces brain blood oxygen level dependent (BOLD) response during exposure to alcohol cues, during a task-based fMRI scan. We will also investigate the effects of PF-05190457 on food craving as well as on food choices using a virtual buffet experimental procedure. All these outcomes will be assessed in the inpatient Unit at the NIH Clinical Center (CC). After the inpatient portion of the protocol, patients will be followed-up as outpatients. During the outpatient phase, patients will be offered motivational interviewing and video feedback to explore the effects of this intervention, compared to supportive counseling, on maintaining motivation for alcohol abstinence and inform future studies where medications like PF-05190457 and behavioral treatments may be combined. The outpatient phase is optional for treatment seeking and nontreatment seeking participants.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male or female individuals 18-70 years old (inclusive)
* Current Alcohol Use Disorder (AUD) by DSM-5 criteria based on the SCID
* Most recent urine drug test for illegal drugs of abuse is negative
* Most recent Clinical Institute Withdrawal Assessment for Alcohol - revised (CIWA-Ar) score is less than or equal to 8
* Heart rate less than or equal to 100 on two separate measurements, both assessed after CIWA-Ar score is less than or equal to 8
* Female subjects must be of non childbearing potential as defined by at least one of the following criteria:

  a) Females 45-70 years old, who are menopausal, defined as follow:

  i) Females who are between 45-55 years old: they will be considered menopausal if they satisfy all the following three requirements during screening: 1) they are in amenorrhea, defined as absence of menstruation for the previous 12 months; 2) they have a negative urine pregnancy test; and 3) they have a serum FSH level within the laboratory s reference range for postmenopausal females.

ii) Females who are between 56-70 years old: they will be considered menopausal if they are in amenorrhea, defined as absence of menstruation for the previous 12 months before screening.

OR

b) Females 21-70 years old, who have a documented hysterectomy and/or bilateral oophorectomy.

All other female subjects (including females with tubal ligations and females that do NOT have a documented hysterectomy) will be considered to be of childbearing potential.

* Male subjects must use one of the following methods of contraception from the first dose of study medication and until 28 days after dosing (given that it is unknown whether the effects of this drug can cause birth defects):

  1. Abstinence.
  2. A condom AND one of the following:

     * Vasectomy for more than 6 months.
     * Female partner who meets one of the following conditions:

       1. Has had a tubal ligation, hysterectomy, or bilateral oophorectomy;
       2. Is post menopausal;
       3. Uses one of the following forms of contraception:

          Copper or hormonal containing IUD;

          Spermicidal foam/gel/film/cream/suppository;

          Diaphragm with spermicide;

          Oral contraceptive;

          Injectable progesterone;

          Subdermal implant.

          EXCLUSION CRITERIA:
* Lifetime clinical diagnosis of schizophrenia or bipolar disorder
* EKG with QTc > 450 msec as determined by the Fridericia formulas.
* BMI less than or equal to 18.5 kg/M(2) or anorexia
* BMI greater than or equal to 40 kg/m(2)
* History of epilepsy and/or seizures

NOTE: individuals who have a history of alcohol withdrawal seizures may be in the study as long as they have been abstinent from alcohol for at least 2 weeks prior to consent and during that period of abstinence, there were no seizure episodes (otherwise, participant remains not eligible).

* Most recent blood tests show creatinine greater than or equal to 2 mg/dL, AST or ALT > 3 times the upper normal limit, hemoglobin <10.5 g/dl
* Subjects who have diabetes and/or are treated with any drug with glucose lowering properties such as sulfonylurea, insulin, metformin, thiazolidinediones (TZD), Dipeptidyl peptidase-4 (DPP4) inhibitors, or Glucagon-like peptide-1(GLP-1)agonists (due to the glucose-lowering properties of PF-05190457 observed in healthy volunteers)
* Exclusionary Medications:

  * A. Naltrexone, acamprosate, alcohol dehydrogenase inhibitors, topiramate, gabapentin, ondansetron, benzodiazepines, baclofen, drugs that are known to prolong the QTc interval and barbiturates as well as hormone replacement therapy; medications and dietary/herbal supplements (like St. John's wort) that interact with Cytochrome P450 3A4. Patients who take these medications may be enrolled in the study only if the potentially interacting medication has been stopped for a period of at least 5 half-lives of the interacting medication before PF-05190457 administration. Patients who take these medications on an as needed (PRN) schedule or take

the medication as a one-time dose as part of a medical procedure or a diagnostic test, for example, may not have to wait the 5 half-lives period of time before enrollment; this will be evaluated on a case by case basis by the MAI and/or PI, based on the specific pharmacological properties of the medication.

* Unable to pass a finger rub hearing test
* Vision is unable to be corrected to (Snellen) 20/100
* Clinically-significant history of motion or car sickness, or history of vestibular disorders
* Any other reason or clinical condition for which the PI or the MAI will consider unsafe for a possible participant to participate in this study

EXCLUSION CRITERIA FOR fMRI ONLY:

* Have contraindications for brain fMRI, as determined by the NIAAA MRI Safety screening form (conducted under the 14-AA-0181 Screening Protocol)
* Colorblindness (this would prevent subject from completing the Stroop task) using the Ishihara Test for Color Deficiency, Concise Edition, 2014.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Leggio, M.D., PhD, Principal Investigator — National Institute on Drug Abuse (NIDA); National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Tyler RE, Pfaff RK, Khan RMN, Loften A, Zurick R, Zeng Y, Arisa OT, Harvey C, Akhlaghi F, Figg WD, Farokhnia M, Leggio L. Pharmacokinetic and pharmacodynamic results from a randomized controlled study with the growth hormone secretagogue receptor blocker PF-5190457 in recently abstinent patients with alcohol use disorder. Int J Neuropsychopharmacol. 2026 Feb 2;29(2):pyaf081. doi: 10.1093/ijnp/pyaf081. PMID 41474196
- [Derived] Faulkner ML, Farokhnia M, Lee MR, Farinelli L, Browning BD, Abshire K, Daurio AM, Munjal V, Deschaine SL, Boukabara SR, Fortney C, Sherman G, Schwandt M, Akhlaghi F, Momenan R, Ross TJ, Persky S, Leggio L. A randomized, double-blind, placebo-controlled study of a GHSR blocker in people with alcohol use disorder. JCI Insight. 2024 Dec 20;9(24):e182331. doi: 10.1172/jci.insight.182331. PMID 39704175
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-AA-0080.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 42 consented participants, 4 participants did not start the study due to screen failure, and 1 did not start the study due to organization issue.
Period: Phase 1
Arm/Group | PF-05190457, Then Placebo | Placebo, Then PF-05190457
Started | 18 | 19
Completed | 17 | 16
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 0 | 1
Period: Washout Period
Arm/Group | PF-05190457, Then Placebo | Placebo, Then PF-05190457
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0
Period: Phase 2
Arm/Group | PF-05190457, Then Placebo | Placebo, Then PF-05190457
Started | 17 | 16
Completed | 16 | 14
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-05190457, Then Placebo | Placebo, Then PF-05190457 | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 19 | 36
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 10 | 17 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 18 | 35
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 8 | 12 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Cue-elicited Craving Assessed in a "Bar-like" Laboratory
Description: Alcohol cue elicited craving was measured using the Alcohol Urges Questionnaire (AUQ). The AUQ is an 8-item self-administered instrument that assesses craving for alcohol among alcohol users in the current context (i.e., right now). The score ranges from 8 (lowest craving value) to 56 (highest craving value).
Time Frame: 96 minutes
Population: The analyses included those participants who completed the entire Cue Reactivity Procedure. 2 participants were not included in the final analysis - 1 for data quality issues and 1 for not completing the entire Cue Reactivity Procedure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- PF-05190457: Participants with alcohol use disorder received PF-05190457 100 mg twice a day for a maximum of 14 days
- Placebo: Participants with alcohol use disorder received placebo twice a day for a maximum of 14 days
Arm/Group | PF-05190457 | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale | 15.52 (1.19) | 15.88 (1.095)

2. Secondary Outcome: Food Choices in a "Virtual Buffet" Conducted in a Virtual Reality Context.
Description: Food choice was assessed by calculating the total of number of calories for a meal selected in a virtual buffet environment. Calories were adjusted for the size of items in the virtual reality environment.
Time Frame: 40 minutes
Population: The analyses included those participants who completed the entire Virtual Reality Procedure. 1 participant was not included in the final analysis due to data quality issues.
Measure: Least Squares Mean (Standard Error); unit: Adjusted calorie count
Arm/Group | PF-05190457 | Placebo
Number analyzed (Participants) | 29 | 29
Adjusted calorie count | 713.6 (39.13) | 848.4 (87.51)

ADVERSE EVENTS:
Time Frame: 35 days
Description: Adverse events were monitored during clinical admission
Arm/Group | PF-05190457 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 13/37 | 15/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-05190457 (N=37) | Placebo (N=37)
Hordeolum (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 5 (7) | 6 (8)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Increased appetite (Metabolism and nutrition disorders) | 3 (3) | 4 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 5 (8)
Insomnia (Nervous system disorders) | 3 (3) | 0 (0)
Lethargy (Nervous system disorders) | 11 (20) | 9 (16)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 1 (1)
Euphoric mood (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of the study due to the COVID-19 pandemic resulted in a smaller number of participants analyzed, compared to the planned sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT02707055/Prot_SAP_000.pdf